CLINICAL TRIAL: NCT00805545
Title: The Timing of Antibiotic Prophylaxis for Cesarean Delivery
Brief Title: Timing of Antibiotic Prophylaxis for Cesarean Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C/S- Antibiotics
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-03

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Group of patients that will receive antibiotics 30-60 minutes prior to incision
  Interventions: Drug: Antibiotic
- B (Active Comparator): Group of patients that will receive antibiotics immediately after clamping the umbilical cord
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — Cefazolin 1gm Intravenously and Azithromycin 500mg Intravenously
  Arms: A
Drug: Antibiotic — Cefazolin 1gm Intravenously and Azithromycin 500mg Intravenously
  Arms: B

SUMMARY:
The current standard of care to prevent post partum infectious morbidities is to administer antibiotic prophylaxis to all women undergoing a cesarean delivery. The general practice is to administer the antibiotic immediately after the umbilical cord is clamped. This study will compare the incidence of post partum infectious morbidities when the extended spectrum prophylaxis given before the incision time vs. the time of cord clamp.

DETAILED DESCRIPTION:
Some studies suggest that administering the antibiotics prior to skin incision decrease the incidence of post partum infectious morbidities without increasing the risks to the baby from the exposure to the antibiotics. Our investigation will validate these findings in a larger series of patients. We will be conducting a prospective controlled randomized trial that will compare both methods of antibiotic prophylaxis. All patients undergoing cesarean delivery will be eligible except for the patients with the diagnosis of chorioamnionitis. One group will receive Cefazolin 1gm intravenous + Azithromycin 500mg intravenous 30-60 minutes prior to incision. The second group will receive the same antibiotics immediately after cord clamp. The primary outcomes will be endometritis, wound infection, neonatal sepsis evaluations, proven cases of neonatal infection. Secondary outcomes will be patients that required post procedure antibiotics, the duration of treatment for mother and neonate and the pattern of antibiotic resistance in microorganisms isolated and characteristics of the neonatal bowel flora.

ELIGIBILITY:
Inclusion Criteria:

* All Patients undergoing cesarean delivery

Exclusion Criteria:

* Patients diagnosed with chorioamnionitis at the time of decision
* Patients that require an emergency cesarean delivery
* Patients that decline participating on the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Duff, M.D., Principal Investigator — Obstetrics and Gynecology; Lorna Rodriguez, M.D., Principal Investigator — Obstetrics and Gynecology
Locations (1):
- Shands Hospital, Gainesville, Florida, United States

REFERENCES:
- [Background] Duff P. Prophylactic antibiotics for cesarean delivery: a simple cost-effective strategy for prevention of postoperative morbidity. Am J Obstet Gynecol. 1987 Oct;157(4 Pt 1):794-8. doi: 10.1016/s0002-9378(87)80057-1. PMID 3118716
- [Background] Tita AT, Hauth JC, Grimes A, Owen J, Stamm AM, Andrews WW. Decreasing incidence of postcesarean endometritis with extended-spectrum antibiotic prophylaxis. Obstet Gynecol. 2008 Jan;111(1):51-6. doi: 10.1097/01.AOG.0000295868.43851.39. PMID 18165392
- [Background] Burke JF. The effective period of preventive antibiotic action in experimental incisions and dermal lesions. Surgery. 1961 Jul;50:161-8. PMID 16722001
- [Background] Sullivan SA, Smith T, Chang E, Hulsey T, Vandorsten JP, Soper D. Administration of cefazolin prior to skin incision is superior to cefazolin at cord clamping in preventing postcesarean infectious morbidity: a randomized, controlled trial. Am J Obstet Gynecol. 2007 May;196(5):455.e1-5. doi: 10.1016/j.ajog.2007.03.022. PMID 17466699
- [Background] Gordon HR, Phelps D, Blanchard K. Prophylactic cesarean section antibiotics: maternal and neonatal morbidity before or after cord clamping. Obstet Gynecol. 1979 Feb;53(2):151-6. PMID 418966
- [Background] Cunningham FG, Leveno KJ, DePalma RT, Roark M, Rosenfeld CR. Perioperative antimicrobials for cesarean delivery: before or after cord clamping? Obstet Gynecol. 1983 Aug;62(2):151-4. PMID 6866355
- [Background] Thigpen BD, Hood WA, Chauhan S, Bufkin L, Bofill J, Magann E, Morrison JC. Timing of prophylactic antibiotic administration in the uninfected laboring gravida: a randomized clinical trial. Am J Obstet Gynecol. 2005 Jun;192(6):1864-8; discussion 1868-71. doi: 10.1016/j.ajog.2004.12.063. PMID 15970833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from November 1, 2008 through November 30, 2009 on the Labor and Delivery unit at the University of Florida.
Pre-assignment Details: We used computer generated random numbers to assign patients to the two groups. Patients were excluded from the study if they were allergic to either of the study drugs or if they had evidence of infection prior to surgery.
Groups:
- Preoperative Antibiotics: Group of patients that will receive antibiotics 30-60 minutes prior to incision
- Post Cord-clamping Antibiotics: Group of patients that will receive antibiotics immediately after clamping the umbilical cord
Period: Overall Study
Arm/Group | Preoperative Antibiotics | Post Cord-clamping Antibiotics
Started | 200 | 200
Completed | 194 | 197
Not Completed | 6 | 3
Not completed — Protocol Violation | 3 | 2
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative Antibiotics | Post Cord-clamping Antibiotics | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 200 | 200 | 400
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.04 (6.6) | 28.9 (5.8) | 28.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 200 | 400
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 200 | 200 | 400

OUTCOME MEASURES:

1. Primary Outcome: Endometritis and Wound Infection
Description: In non-pregnant patients having certain types of surgery with a high risk of infection, prophylactic antibiotics are routinely administered before the surgical procedure begins to ensure that a high level of antibiotic is present in tissue prior to the time that maximum bacterial contamination occurs. However, there has been concern about exposing the fetus in utero to antibiotics. The question to be addressed was whether preoperative antibiotics (as opposed to antibiotics administered after clamping of the umbilical cord) benefitted the mother without increasing risk for the baby.
Time Frame: Patients were followed from the time of surgery until 6 weeks postpartum.
Population: All 194 patients who received preoperative antibiotics and who completed the study were analyzed. All 197 patients who received post-cord clamping antibiotics and who completed the study were analyzed.
Measure: Number (95% Confidence Interval); unit: patients infected
Arm/Group | Preoperative Antibiotics | Post Cord-clamping Antibiotics
Number analyzed (Participants) | 194 | 197
patients infected | 6 [0.142 to 7.28] | 4 [0.372 to 11.34]

ADVERSE EVENTS:
Time Frame: 1 year
Description: We evaluated the frequency of endometritis and wound infection in study patients. We also assessed patients for possible adverse effects related to administration of prophylatic antibiotics.
Arm/Group | Preoperative Antibiotics | Post Cord-clamping Antibiotics
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 6/200 | 4/200
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoperative Antibiotics (N=200) | Post Cord-clamping Antibiotics (N=200)
Endometritis and wound infection (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 4 (4) — We evaluated the frequency of postoperative endometritis and wound infection in the patients who received prophylactic antibiotics.

LIMITATIONS AND CAVEATS:
There were no limitations to the study. No technical problems occurred during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes